CLINICAL TRIAL: NCT04721652
Title: Fluid Intake After Hemodialysis: Investigating the Relationship Between Time and Weight Gain During the Interdialytic Interval
Brief Title: Fluid Intake After Hemodialysis
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Principal Investigator, Director of The Lilibeth Caberto Kidney Clinical Research Unit, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 117983
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Interdialytic Weight Gain
Keywords: Hemodialysis; Interdialytic Weight Gain; Thirst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hemodialysis Patients (nondiabetic): Nondiabetic adult hemodialysis patients

SUMMARY:
Interdialytic weight gain determines how much fluid (ultrafiltration) has to be removed during each hemodialysis session. High ultrafiltration volumes stress the organism and lead to a higher risk of death. Thirst is the main driving factor of interdialytic weight gain, and thirst is mainly driven by salt intake, molecules that increase blood tonicity (such as sugar in diabetics) and fluid loss (such as in dehydration and blood loss). It has been speculated that fluid loss during hemodialysis could increase the sense of thirst immediately following dialysis, but this statement requires further evidence.

DETAILED DESCRIPTION:
Overview: In this observational study, we will have a sample of approximately 20 patients on chronic thrice weekly HD self-monitor their weight gain and blood pressure during the interdialytic intervals for one week. Demographics, anthropometrics, HD prescription and treatment information will be recorded. Study participants will complete four questionnaires at the first study visit and will then be provided medical grade scales and a blood pressure monitor, and will be asked to prospectively record weight changes and blood pressure at home four times a day for one week using a logbook.

Patients with significant residual urinary volume and diabetes mellitus will not be recruited, the latter to remove the bias of blood glucose in determining osmotic thirst.

Home Body Weight Monitoring Study participants will be asked to perform daily home body weight monitoring for the duration of the whole study with medical grade scales. Study participants will be asked to monitor their body weight four times per day: upon waking up, between 12:00 and 2:00 pm, between 6:00 and 8:00 pm and at bedtime. Participants will be asked to wear similar clothing for all measurements. Monitoring will start after the first HD session of the week until the first HD session of the following week.

Home Blood Pressure Monitoring Study participants will be asked to perform daily home blood pressure monitoring for the duration of the whole study with a validated, automated device. Participants with an arteriovenous fistula or graft will be asked to measure blood pressure on the arm without the arteriovenous fistula or graft. Study participants will be asked to monitor blood pressure four times per day, concomitantly with their body weight. Study participants will be asked to record three consecutive blood pressure measurements in a sitting position, after 5 minutes of rest in a quiet room. Monitoring will start after the first HD session of the week until the first HD session of the following week.

Daily Reminders Study participants will be given the option to receive a daily reminder phone call for the duration of the whole study, to encourage compliance to the self-monitoring procedures and to encourage reproducibility (e.g. by wearing similar clothing at each measurement) to weighing procedures. The phone calls will be made from an in-hospital office phone by either the research coordinators or the Ph.D. student attached to this study, following a script. Participants can decline the option of receiving daily reminders.

Scored Sodium Questionnaire Dietary sodium intake will be estimated with the Scored Sodium Questionnaire (SSQ)12 on the first study visit, a 10-item food frequency questionnaire to screen for high sodium intake in CKD. A cut-off value of 65 will be used to identify patients with high sodium intake.

Dialysis Thirst Inventory The Dialysis Thirst Inventory (DTI) is a questionnaire developed by Bots et al.13 It is a seven items questionnaire that quantifies the perception of thirst. Each item has a five-point Likert type scale (never = 1, to very often = 5). The scores are summed and provide a DTI score ranging from 7 (no thirst) to 35 (very thirsty). The items are the following: (1) Thirst is a problem for me. (2) I am thirsty during the day. (3) I am thirsty during the night. (4) My social life is influenced because of my thirst feelings; (5) I'm thirsty before dialysis. (6) I am thirsty during dialysis. (7) I am thirsty after dialysis. This questionnaire will be administered on the first study visit.

Xerostomia Inventory The validated Xerostomia Inventory (XI) consists of 11 items, each with a five-point Likert type scale (never=1, to very often=5) to evaluate xerostomia, that is a feeling of dry mouth.14 Examples of items from the XI are "My mouth feels dry...", "I have difficulty in eating dry foods..." and "I sip liquids to aid in swallowing food." The responses to the 11 items result in an individual XI score for each participant that can range from 11 (no dry mouth) to 55 (extremely dry mouth). This questionnaire will be administered on the first study visit.

Minutes to Recovery after HD This is a clinically validated, simple question, as published by Lindsay et al.15 The question is: "How long does it take you to recover from a dialysis session?", to which participants are free to respond by providing exact times to approximate estimates such as "half a day". The final answer will be converted to minutes for analysis purposes. Responses to this question were reported to be highly reproducible over time and correlated with several quality of life questionnaires, mainly pointing towards physical wellbeing rather than mental health. Furthermore, this measure was sensitive enough to show differences in recovery time between different HD prescriptions (standard vs daily vs nocturnal HD). This question will be administered on the first study visit.

Urine collection When applicable, participants will be asked to collect and record their urine volume on the last day of the long interdialytic interval (Sunday for Monday-Wednesday-Friday patients, Monday for Tuesday-Thursday-Saturday patients). Participants will be provided a disposable urine collection container for this purpose. After completing the collection and recording the total urine volume, the participants will dispose of the urine themselves.

Concomitant Medications Throughout the study, all participants will continue to take all medications as prescribed by their clinical care team and will follow any changes to their medication as seen fit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Thrice weekly maintenance hemodialysis
* Willing and able to provide written informed consent

Exclusion Criteria:

* Diabetes Mellitus
* Residual Urinary Volume > 500 ml/day
* Being able to self-monitor one's body weight and blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this observational study, we will have a sample of approximately 20 patients on chronic thrice weekly HD self-monitor their weight gain and blood pressure during the interdialytic intervals for one week. Demographics, anthropometrics, HD prescription and treatment information will be recorded. Study participants will complete four questionnaires at the first study visit and will then be provided medical grade scales and a blood pressure monitor, and will be asked to prospectively record weight changes and blood pressure at home four times a day for one week using a logbook.
  Patients with significant residual urinary volume and diabetes mellitus will not be recruited, the latter to remove the bias of blood glucose in determining osmotic thirst.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
T50%IDWG | Up to one week
  Time to achieve ≥50% cumulative interdialytic weight gain (T50%IDWG) from the last hemodialysis treatment
Cumulative IDWG% curve | Up to one week
  Shape of cumulative interdialytic weight gain curve (linear vs nonlinear)

SECONDARY OUTCOMES:
Correlations of T50%IDWG | One week, Interdialytic intervals
  Correlation between T50%IDWG with comorbid heart failure, ultrafiltration volume, ultrafiltration rate, intradialytic hypotension, minutes to recovery after hemodialysis, dialysate sodium concentration, scored sodium questionnaire, dialysis thirst inventory, xerostomia inventory.
Correlations of Nighttime cumulative %IDWG | One week, Interdialytic intervals
  Correlation between Nighttime cumulative %IDWG with comorbid heart failure, ultrafiltration volume, ultrafiltration rate, intradialytic hypotension, minutes to recovery after hemodialysis, dialysate sodium concentration, scored sodium questionnaire, dialysis thirst inventory, xerostomia inventory.
Comparisons between IDWG% curves | One week, Interdialytic intervals
  Compare prevalence in comorbid heart failure, ultrafiltration volume, ultrafiltration rate, intradialytic hypotension minutes to recovery after hemodialysis, dialysate sodium concentration, scored sodium questionnaire, dialysis thirst inventory, xerostomia inventory in patients with linear vs nonlinear cumulative interdialytic weight gain curve
Daytime vs Nighttime cumulative IDWG% | One week, Interdialytic intervals
  Comparison between Daytime vs Nighttime cumulative interdialytic weight gain %

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. McIntyre, MD, PhD, Principal Investigator — London Health Sciences Centre, Western University
Locations (2):
- Canada (2):
  - Adam Linton Unit, London, Ontario
  - Westmount Kidney Care Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No